CLINICAL TRIAL: NCT01177488
Title: Innovative Service Delivery for Secondary Prevention of PTSD in At-Risk OIF-OEF Service Men and Women
Brief Title: Innovative Service Delivery for Secondary Prevention of PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charleston Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DoD Acierno
Record Dates: First submitted 2010-04-12; First posted 2010-08-09 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: PTSD
Keywords: Military; Health Service Delivery; Behavioral Symptoms; Telepsychology; Behavioral Activation; Exposure Therapy; Veterans; Telemedicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BATE-T (Experimental): Behavioral Activation Therapeutic Exposure done while the patient is at home via videoconferencing technology
  Interventions: Behavioral: Behavioral Activation Therapeutic Exposure (BATE)
- BATE-IP (Active Comparator): Behavioral Activation Therapeutic Exposure done in the therapist's office
  Interventions: Behavioral: Behavioral Activation Therapeutic Exposure (BATE)

INTERVENTIONS:
Behavioral: Behavioral Activation Therapeutic Exposure (BATE) — This intervention combines Behavior Activation Therapy and Exposure Therapy to treat PTSD symptoms.

SUMMARY:
The purpose of this study is to determine whether therapy for Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) veterans with Post-traumatic Stress Disorder (PTSD) symptoms can be delivered effectively using videoconferencing technology ("telepsychology"), which allows a therapist and patient who are not in the same room as one another to communicate.

DETAILED DESCRIPTION:
OIF and OEF service men and women exposed to high levels of violence are at risk for developing mental health disorders including Post-traumatic Stress Disorder (PTSD) and Major Depressive Disorder (MDD). Even those with less severe symptoms who fail to meet diagnostic criteria for a mental health disorder may struggle to return to pre-deployment functioning. Studies suggest that a significant percentage of veterans may suffer from "subthreshold" PTSD; although their symptom presentation is less severe, these veterans experience emotional distress and reduced quality of life.

Given that Veterans Affairs (VA) mental-health service providers are faced with the important and challenging task of alleviating the emotional suffering of our service men and women while staying within budget confines, we need effective, practical, evidence-based treatments that can be delivered in an expedient and cost-effective manner. Thus, the current project has two primary objectives: 1) to develop, implement, and evaluate a treatment program (Behavioral Activation and Therapeutic Exposure, BATE) for OIF and OEF veterans with PTSD symptoms, and 2) to determine whether or not this program delivered via telepsychology will be as effective as in-person treatment. Secondary objectives include determining: 1) which treatment modality is more effective in terms of process variables (e.g., treatment satisfaction, session attendance), 2) which treatment modality is more cost-effective, and 3) whether treatment effects differ across race and gender. Study participants will be randomized to two treatment conditions, BATE delivered via telepsychology (BATE-T) and BATE delivered in-person (BATE-IP).

The current treatment protocol is based on two, research-supported therapeutic rationales, Behavioral Activation (BA) and Therapeutic Exposure (TE). Briefly, the treatment aims to increase the participant's engagement in healthy activities (i.e., activities that are naturally reinforcing and promote the participant's life values) and exposure activities (i.e., activities that target specific PTSD symptoms such as avoidance and hyperarousal). Treatment will be implemented in eight, one and half hour sessions. Although research supports the effectiveness of behavior- and exposure-based treatments for trauma-related mental health problems, a potential risk for any counseling program that targets avoidance symptoms is a temporary increase in emotional distress. Therapists will inform participants that this is a normal "side effect" of treatment. However, over the course of treatment should a participant's emotional distress rise to a level above what can be handled via outpatient counseling, the participant will be removed from the study and appropriate referrals will be made.

The anticipated duration of this study is four years. Based on results of the study, we will finalize the treatment manual. In terms of clinical applicability, we plan to present study findings at conferences and disseminate the treatment manual to VA mental health service providers in approximately four to five years. Study findings will address important gaps in the PTSD literature, yielding several contributions to the field. First, to the extent that BATE effectively reduces symptom severity, this investigational treatment may benefit individual OIF/OEF service men and women by alleviating emotional suffering and improving quality of life. Second, to the extent that BATE prevents the development of full-blown PTSD in subclinical military personnel, this investigational treatment may reduce attrition from the military due to untreated mental health problems. Third, only a small percentage of those who might benefit from counseling actually seek services due to barriers associated with traditional service delivery practices such as geographic distance from the VA hospital and stigma of psychological treatment. Thus, as telemedicine has been shown to circumvent these barriers to care, the current project has the potential to reach an otherwise underserved population: subclinical OIF and OEF service men and women who may be reluctant to seek care. Fourth, to the extent that BATE-T produces results comparable to BATE-IP, this study may potentially identify a cost-effective alternative to in-person treatment thereby reducing post-service treatment costs to VA's.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be OIF/OEF military personnel,
* age 21 and above, and
* with symptoms of posttraumatic stress disorder (PTSD) assigned on the basis of the Clinician Administered PTSD Scale (CAPS) and PTSD Checklist-Military (PCL-M).

Exclusion Criteria:

* Actively psychotic or demented persons,
* individuals with both suicidal ideation and clear intent, and
* individuals meeting criteria for substance dependence will be excluded from participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-03; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The major objective of this study is to determine if Behavioral Activation with Therapeutic Exposure (BATE) delivered via Telemedicine is as effective as BATE In Person. | 1 year
  This is measured in terms of (1) clinical (PTSD and Depression); (2) process (Treatment Satisfaction and Attrition); and (3) economic (Cost) outcomes.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | Baseline
Clinician Administered PTSD Scale (CAPS) | 8 weeks
Clinician Administered PTSD Scale (CAPS) | 3 months
Clinician Administered PTSD Scale (CAPS) | 1 year
The Deployment Risk and Resiliency Inventory (DRRI) | Baseline
PTSD Checklist-Military (PCL-M) | Baseline
PTSD Checklist-Military (PCL-M) | 4 weeks
PTSD Checklist-Military (PCL-M) | 8 weeks
PTSD Checklist-Military (PCL-M) | 3 months
PTSD Checklist-Military (PCL-M) | 1 year
Beck Depression Inventory-II (BDI-II) | Baseline
Beck Depression Inventory-II (BDI-II) | 4 weeks
Beck Depression Inventory-II (BDI-II) | 8 weeks
Beck Depression Inventory-II (BDI-II) | 3 months
Beck Depression Inventory-II (BDI-II) | 1 year
Health Related Functioning: Medical Outcome Study Short Study Forms-36 Health Survey (SF 36) | Baseline
Health Related Functioning: Medical Outcome Study Short Study Forms-36 Health Survey (SF 36) | 4 weeks
Health Related Functioning: Medical Outcome Study Short Study Forms-36 Health Survey (SF 36) | 8 weeks
Health Related Functioning: Medical Outcome Study Short Study Forms-36 Health Survey (SF 36) | 3 months
Health Related Functioning: Medical Outcome Study Short Study Forms-36 Health Survey (SF 36) | 1 year
Charleston Psychiatric Outpatient Satisfaction Scale (CPOSS-VA) | 8 weeks
Service Delivery Perceptions Questionnaire | 8 weeks
Prior Experience with Computer and Audiovisual Technology | Baseline
  Short measure to learn more about participants' prior experience and comfort level with computers and audiovisual technology

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Acierno, PhD, Principal Investigator — VA Office of Research and Development
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph H. Johnson VAMC, Charleston, South Carolina

REFERENCES:
- [Background] Acierno R, Rheingold A, Amstadter A, Kurent J, Amella E, Resnick H, Muzzy W, Lejuez C. Behavioral activation and therapeutic exposure for bereavement in older adults. Am J Hosp Palliat Care. 2012 Feb;29(1):13-25. doi: 10.1177/1049909111411471. Epub 2011 Jun 17. PMID 21685428
- [Background] Gros DF, Price M, Yuen EK, Acierno R. Predictors of completion of exposure therapy in OEF/OIF veterans with posttraumatic stress disorder. Depress Anxiety. 2013 Nov;30(11):1107-13. doi: 10.1002/da.22207. Epub 2013 Oct 21. PMID 24151141
- [Background] Gros DF, Price M, Strachan M, Yuen EK, Milanak ME, Acierno R. Behavioral activation and therapeutic exposure: an investigation of relative symptom changes in PTSD and depression during the course of integrated behavioral activation, situational exposure, and imaginal exposure techniques. Behav Modif. 2012 Jul;36(4):580-99. doi: 10.1177/0145445512448097. Epub 2012 Jun 7. PMID 22679240
- [Background] Gros DF, Strachan M, Ruggiero KJ, Knapp RG, Frueh BC, Egede LE, Lejuez CW, Tuerk PW, Acierno R. Innovative service delivery for secondary prevention of PTSD in at-risk OIF-OEF service men and women. Contemp Clin Trials. 2011 Jan;32(1):122-8. doi: 10.1016/j.cct.2010.10.003. Epub 2010 Oct 14. PMID 20951235
- [Background] Gros DF, Veronee K, Strachan M, Ruggiero KJ, Acierno R. Managing suicidality in home-based telehealth. J Telemed Telecare. 2011;17(6):332-5. doi: 10.1258/jtt.2011.101207. Epub 2011 Aug 15. PMID 21844180
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Price M, Gros DF, Strachan M, Ruggiero KJ, Acierno R. Combat experiences, pre-deployment training, and outcome of exposure therapy for post-traumatic stress disorder in Operation Enduring Freedom/Operation Iraqi Freedom veterans. Clin Psychol Psychother. 2013 Jul-Aug;20(4):277-85. doi: 10.1002/cpp.1768. Epub 2012 Jan 18. PMID 22253233
- [Background] Price M, Gros DF, Strachan M, Ruggiero KJ, Acierno R. The Role of Social Support in Exposure Therapy for Operation Iraqi Freedom/Operation Enduring Freedom Veterans: A Preliminary Investigation. Psychol Trauma. 2013 Jan 1;5(1):93-100. doi: 10.1037/a0026244. PMID 23869250
- [Background] Strachan M, Gros DF, Ruggiero KJ, Lejuez CW, Acierno R. An integrated approach to delivering exposure-based treatment for symptoms of PTSD and depression in OIF/OEF veterans: preliminary findings. Behav Ther. 2012 Sep;43(3):560-9. doi: 10.1016/j.beth.2011.03.003. Epub 2011 May 24. PMID 22697444
- [Background] Strachan M, Gros DF, Yuen E, Ruggiero KJ, Foa EB, Acierno R. Home-based telehealth to deliver evidence-based psychotherapy in veterans with PTSD. Contemp Clin Trials. 2012 Mar;33(2):402-9. doi: 10.1016/j.cct.2011.11.007. Epub 2011 Nov 11. PMID 22101225